CLINICAL TRIAL: NCT03979950
Title: Contraception for Solid Organ Transplant Patients: Utilizing Social Media
Status: Completed | Type: Observational
Sponsor: University of California, San Diego (Other)
Collaborators: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Sheila Mody, Assistant Professor, University of California, San Diego
Other Study IDs: 170592X
Record Dates: First submitted 2018-03-13; First posted 2019-06-10 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Contraception; Contraception Behavior; Contraceptive Usage; Reproductive Health
Keywords: organ transplant
MeSH Terms: conditions — Contraception Behavior | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Survey — Solid Organ Transplant patients will be recruited via social media. Co-investigators will reach out to the administrators of various social media networks to share information regarding the study with their networks on our behalf. Potential participants who are interested in participating, can then follow the link to the online survey tool, which includes the participant demographic information (age, ethnicity and highest level of education) and questionnaire. The questionnaire is 30 questions long and takes approximately 15 minutes to complete. This questionnaire will be a single, cross-sectional survey. No personal information will be documented on the questionnaire. All responses will be anonymous. Participants will be recruited for 6 months.

SUMMARY:
The purpose of this study is to use an electronic survey to explore Solid Organ Transplant patients' contraceptive knowledge and counseling. The results from this survey will be used to help identify awareness gaps to potentially develop targeted interventions for comprehensive education.

DETAILED DESCRIPTION:
According to data from the U.S. Organ Procurement and Transplantation Network, 10,804 women received organ transplants in 2011. Of these women, 3896 (36%) were between the ages of 18 and 49. Women of reproductive age make up a significant part of the transplant recipient population, so pregnancy in these immunocompromised patients is a concern. The incidence of unwanted pregnancy (a subset of unintended pregnancies) among female kidney transplant recipients is 48%, while the national incidence is 25%. The American Society of Transplantation (AST) has come to a consensus that gestations in organ transplant patients be considered high risk and be managed by both transplant physicians and high-risk pregnancy specialists. Pregnancies after organ transplantation have a high incidence of low birth weight (less than 2.5 kg).

The risks posed to the woman herself, her transplanted organ, and fetus underscore the importance of having health care providers counsel transplant patients on family planning, including return to fertility, contraceptive use, and when pregnancy can be safely considered. Specifically the fetus may be exposed to teratogenic immunosuppressive transplant medications and pregnancy increases the risk for rejection of the transplanted organ. Therefore it is important that women are thoroughly counseled regarding contraceptive effectiveness and safety. Health care providers have a large impact on the reproductive decisions that patients make. In a study done in transplant clinics across the nation, the majority of respondents based their decision on whether to become pregnant on the guidance of the individual transplant physician.

Transplant specialists may not be comfortably providing family planning services directly to patients. The Center for Disease Control and Prevention's United States Medical Eligibility Criteria for Contraceptive Use has specific guidance on the safety of each contraceptive for women undergoing solid organ transplants. However, this guidance is based on limited safety data. This study aims to add to the literature available on this patient population although we are not assessing safety. In addition, this study will identify improvement opportunities to the care provided to transplant patients within our own Health System.

This research study is a unique collaboration between the Departments of Pharmacy, Nephrology, and Reproductive Medicine.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-50 years old, solid organ transplant in the last 5 years, and fluent in English.

Exclusion Criteria:

* Not sexually active with men, history of hysterectomy, history of oophorectomy

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Study Population: Women 18-50 years, solid organ transplant in the last 5 years, and fluent in English.
Sampling Method: Non-Probability Sample
Enrollment: 52 (Actual)
Dates: Start 2018-01-18 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-12-01 (Actual)

PRIMARY OUTCOMES:
Level of knowledge among solid organ transplant patients about contraceptive methods | Three years
  The survey questionnaire asks multiple-choice questions about (1) available contraceptive methods, (2) the safety profile of methods for women with transplant histories, and (3) the teratogenic risks of post-transplant medications.
Quantity of contraceptive counseling for solid organ transplant patients | Three years
  The survey questionnaire asks multiple-choice questions about (1) whether patients received counseling about contraception and (2) if they want more counseling on contraception.
Number of participants counseled on contraception by provider | Three years
  The survey questionnaire asked multiple-choice questions about (1) which, if any, provider(s) counseled them on contraception and (2) from which provider(s), if any, would they prefer to receive contraceptive counseling.

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD, MPH, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Organ Procurement and Transplantation Network. Organ Procurement and Transplantation Network, HRSA, DHHS 9 A.D. November 10. Available from http://optn.transplant.hrsa.gov/.
- [Background] Lessan-Pezeshki M, Ghazizadeh S, Khatami MR, Mahdavi M, Razeghi E, Seifi S, Ahmadi F, Maziar S. Fertility and contraceptive issues after kidney transplantation in women. Transplant Proc. 2004 Jun;36(5):1405-6. doi: 10.1016/j.transproceed.2004.04.090. PMID 15251344
- [Background] McKay DB, Josephson MA, Armenti VT, August P, Coscia LA, Davis CL, Davison JM, Easterling T, Friedman JE, Hou S, Karlix J, Lake KD, Lindheimer M, Matas AJ, Moritz MJ, Riely CA, Ross LF, Scott JR, Wagoner LE, Wrenshall L, Adams PL, Bumgardner GL, Fine RN, Goral S, Krams SM, Martinez OM, Tolkoff-Rubin N, Pavlakis M, Scantlebury V; Women's Health Committee of the American Society of Transplantation. Reproduction and transplantation: report on the AST Consensus Conference on Reproductive Issues and Transplantation. Am J Transplant. 2005 Jul;5(7):1592-9. doi: 10.1111/j.1600-6143.2005.00969.x. PMID 15943616
- [Background] McKay DB, Adams PL, Bumgardner GL, Davis CL, Fine RN, Krams SM, Martinez OM, Murphy B, Pavlakis M, Tolkoff-Rubin N, Sherman MS, Josephson MA. Reproduction and pregnancy in transplant recipients: current practices. Prog Transplant. 2006 Jun;16(2):127-32. doi: 10.1177/152692480601600206. PMID 16789701
- [Background] Centers for Disease Control and Prevention (CDC). U S. Medical Eligibility Criteria for Contraceptive Use, 2010. MMWR Recomm Rep. 2010 Jun 18;59(RR-4):1-86. PMID 20559203
- [Background] Guazzelli CA, Torloni MR, Sanches TF, Barbieri M, Pestana JO. Contraceptive counseling and use among 197 female kidney transplant recipients. Transplantation. 2008 Sep 15;86(5):669-72. doi: 10.1097/TP.0b013e3181817e7d. PMID 18791448
- See also: Centers for Disease Control (CDC) US Medical Eligibility Criteria (US MEC) for Contraceptive Use, 2010 — http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5904a1.htm?s_cid=rr5904a1_e.